CLINICAL TRIAL: NCT07018427
Title: Efficacy and Safety of Sacituzumab Govitecan in Heavily Pretreated Unresectable Locally Advanced, Recurrent, or Metastatic HER2-Negative Breast Cancer: A Multicenter Real-World Study
Brief Title: Real-world Study of Sacituzumab Govitecan Monotherapy or Combination Therapy in Recurrent or Metastatic HER2-negative Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, songguohong, Chief Physician, Deputy Director of the Department, Medical Oncology of Breast Cancer, Peking University Cancer Hospital & Institute
Other Study IDs: RWS119351420
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasms; Triple Negative Breast Cancer; HR+, HER2-, Advanced Breast Cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients received SG: HER2-negative breast cancer patients who received SG treatment in the advanced stage
  Interventions: Drug: Sacituzumab Govitecan Monotherapy or Combination Therapy

INTERVENTIONS:
Drug: Sacituzumab Govitecan Monotherapy or Combination Therapy — The interventions in this study comprised either Sacituzumab Govitecan monotherapy or combination therapy. The specific combination regimens were determined based on real - world clinical practice patterns.
  Other Names: SG

SUMMARY:
This multicenter observational real-world study is planned to enroll 100 patients, divided into two cohorts: the triple-negative breast cancer (TNBC) cohort and the hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer (HR+/HER2- BC) cohort. The study aims to evaluate the efficacy and safety of sacituzumab govetican (SG) monotherapy or combination regimens in patients with unresectable locally advanced, recurrent, or metastatic HER2-negative breast cancer within a real-world context.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Gender Male or female aged 18 years or older.
2. Pathological Diagnosis and Classification Criteria (Must Meet Either Cohort Condition) 2.1 Triple-Negative Breast Cancer (TNBC) Cohort

   Histologically/cytologically confirmed triple-negative breast cancer (TNBC) by pre-SG biopsy/pathology report, with the following criteria:

   HER2-negative: Immunohistochemistry (IHC) score of 0 or 1+; if IHC score is 2+, HER2 negativity must be confirmed by fluorescence in situ hybridization (FISH).

   Estrogen and progesterone receptor-negative: <1% of cells express hormone receptors as determined by IHC.

   Presence of locally advanced, recurrent, or metastatic disease (locally advanced disease must be confirmed by investigators as ineligible for curative resection).

   2.2 Hormone Receptor-Positive/HER2-Negative Breast Cancer (HR+/HER2- BC) Cohort

   Histologically/cytologically confirmed HR+/HER2- breast cancer by pre-SG biopsy/pathology report, with the following criteria:

   HER2-negative: Immunohistochemistry (IHC) score of 0 or 1+; if IHC score is 2+, HER2 negativity must be confirmed by fluorescence in situ hybridization (FISH).

   HR-positive: Hormone receptor positivity (HR, including ER or PR status) is defined as ≥1% cell expression by IHC.

   Presence of locally advanced, recurrent, or metastatic disease (locally advanced disease must be confirmed by investigators as ineligible for curative resection).
3. Treatment Protocol Requirements Planned to receive SG monotherapy or combination therapy.
4. Other Enrollment Criteria Willing to participate in the study, sign the informed consent form, and demonstrate good compliance.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Known allergy to sacituzumab govitecan (SG) or any of its components.
3. History of other malignancies, except the following:

   Cured basal cell carcinoma, squamous cell skin carcinoma, cervical in situ carcinoma, or papillary thyroid carcinoma.

   A second primary cancer that has been completely cured with a tumor-free interval of ≥5 years.

   Other malignancies where the primary tumor source of metastatic foci has been clearly identified by investigators.
4. Diagnosis of other malignancies within the past 5 years
5. Current participation in other interventional clinical studies.
6. Presence of acute or chronic infections, or coexisting serious diseases (such as decompensated heart, lung, liver, or renal failure), assessed by investigators as incompatible with tolerating the study treatment.
7. Mental illness or psychiatric disorders leading to poor compliance, inability to cooperate with the study, or inability to describe treatment responses.
8. Modification of the treatment regimen after SG administration for reasons other than disease progression.
9. Any other circumstances deemed by investigators as likely to interfere with study evaluation, affect subject safety, or render the patient unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable locally advanced, recurrent, or metastatic HER2-negative breast cancer received SG
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Real world progression free survival (rwPFS) | 12 months after the last patient was enrolled
  The time interval from the date of Sacituzumab Govitecan initiation until date of progressive disease (PD) or death from any causes, whichever occurred first.

SECONDARY OUTCOMES:
Real world objective response rate (rwORR) | approximately up to 24 weeks from the initiation of the study treatment.
  The percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Real world overall survival (rwOS) | up to 48 months from the initiation of the study treatment.
  Time from initiation of SG monotherapy or combination therapy to death from any cause
Number of patients with adverse events | approximately up to 68 weeks from the initiation of the treatment.
  Adverse events were assessed during study treatment and at follow-up visits

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No